CLINICAL TRIAL: NCT06859775
Title: Open-label, Multicenter Phase Ib/II Clinical Study of Injectable SHR-A1811 in Combination Regimens for the Treatment of Recurrent or Metastatic Cervical Cancer
Brief Title: SHR-A1811 Combination Regimen for the Treatment of Recurrent or Metastatic Cervical Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-216-CC
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Recurrent or Metastatic Cervical Cancer
MeSH Terms: conditions — Recurrence; Uterine Cervical Neoplasms | interventions — Bevacizumab; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment cohort 1 (Experimental)
  Interventions: Drug: SHR-A1811; Drug: Adebelimab injection; Drug: Bevacizumab injection
- Treatment cohort 2 (Experimental)
  Interventions: Drug: SHR-A1811; Drug: Adebelimab injection; Drug: Bevacizumab injection; Drug: SHR-8068
- Treatment cohort 3 (Experimental)
  Interventions: Drug: SHR-A1811; Drug: Adebelimab injection; Drug: Bevacizumab injection; Drug: SHR-8068; Drug: Cisplatin injection; Drug: Carboplatin injection

INTERVENTIONS:
Drug: SHR-A1811 — SHR-A1811 injection.
Drug: Adebelimab injection — Adebelimab injection.
Drug: Bevacizumab injection — Bevacizumab injection.
Drug: SHR-8068 — SHR-8068 injection.
  Arms: Treatment cohort 2; Treatment cohort 3
Drug: Cisplatin injection — Cisplatin injection.
  Arms: Treatment cohort 3
Drug: Carboplatin injection — Carboplatin injection.
  Arms: Treatment cohort 3

SUMMARY:
This study is a multicentre, open-label, dose-finding/efficacy-expanding phase Ib/II clinical trial to evaluate the tolerability, safety, pharmacokinetic profile and immunogenicity of SHR-A1811 combination regimen in the treatment of recurrent or metastatic cervical cancer and to preliminarily evaluate the efficacy of SHR-A1811 combination regimen for recurrent or metastatic cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily join this study, sign the informed consent form, have good compliance and be able to cooperate with the follow-up.
2. Female, aged 18-75 years old.
3. Expected survival ≥ 12 weeks.
4. Normal function of vital organs.
5. Female subjects of childbearing potential must have a negative serum HCG test within 7 days prior to the first dose and must be non-lactating.
6. Female subjects must agree to comply with contraceptive requirements from signing the informed consent form to 7 months after the last dose of the investigational drug.

Exclusion Criteria:

1. Previous or concomitant other malignancies.
2. Severe bone damage caused by bone metastasis from tumours.
3. Presence of active autoimmune disease or history of autoimmune disease with possible recurrence.
4. Those with active tuberculosis.
5. Concomitant poorly controlled or severe cardiovascular disease.
6. Occurrence of arteriovenous thrombotic events within 6 months prior to the first dose.
7. Presence of gastrointestinal obstruction or presence of symptoms and signs of gastrointestinal obstruction within 6 months prior to the first dose.
8. Subjects who have had a serious infection within 1 month before the first dose.
9. Subjects who have a history of immunodeficiency.
10. As judged by the investigator, there are other factors that may affect the results of the study or cause the study to be forced to terminate halfway.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Grade≥3 drug-related adverse events (TRAEs). | Up to 3 years.
Grade≥3 drug-related serious adverse events (TRAEs). | Up to 3 years.
Objective response rate (ORR). | Up to 3 years.

SECONDARY OUTCOMES:
Duration of response (DOR). | Up to 3 years.
Disease control rate (DCR). | Up to 3 years.
Progression-free survival (PFS). | Up to 3 years.
Overall survival (OS). | Up to 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided